CLINICAL TRIAL: NCT06855394
Title: Impact of CYP2C19 Gene Polymorphism on Long-term Major Adverse Cardiac and Vascular Events
Brief Title: Genetic Testing of CYP2C19 in Prognostic Evaluation of Long-Term Major Adverse Cardiac and Vascular Events
Acronym: UF-GENOTYPE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202302158
Record Dates: First submitted 2025-02-28; First posted 2025-03-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Vascular Disease; Coronary Arterial Disease (CAD); Atherosclerosis of Coronary Artery; Atherosclerosis of Arteries of the Extremities, Unspecified; Heart Diseases; Stroke; Venous Thromboembolic Disease
Keywords: Cardiovascular disease; Atherosclerotic vascular disease; Coronary artery disease; Stroke
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Heart Diseases; Stroke; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buccal swab used to extract DNA for evaluation of specific hepatic cytochrome P450 2C19 alleles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cytochrome P450 2C19 Loss-of-function: Patients carriers of a Cytochrome P450 2C19 loss-of-function allele (i.e., *2 or *3)
- Cytochrome P450 2C19 Non-loss-of-function: Patients without a Cytochrome P450 2C19 loss-of-function allele.

SUMMARY:
Several studies have shown that the efficacy of clopidogrel for secondary prevention of major adverse cardiovascular events (MACE), including acute coronary syndrome, depends on the polymorphism of the CYP2C19 gene. However, studies with large sample sizes and long-term follow-up are missing. Moreover, the impact of this polymorphism on the risk of major adverse limb events (MALE), particularly in patients with peripheral artery disease of the lower limb, is unexplored. Additionally, the impact of CYP2C19 gene polymorphism on clopidogrel effectiveness in preventing recurrent stroke in diverse populations is unknown since most of the data are from Asian ancestry populations. We hypothesize that patients with CYP2C19 gene loss of function alleles are at high risk of MACE and MALE compared to those without loss of function alleles at long-term follow-up. We propose to assess MACE and MALE in a large cohort of patients with available CYP2C19 genotypes treated at the University of Florida Health to evaluate the impact of CYP2C19 gene polymorphisms on the risk of new or recurrent events at long-term follow-up. Our specific aims are Aim 1) to determine the impact of CYP2C19 gene polymorphisms (loss of function alleles vs. non-loss of function alleles) on the risk of MACE (a composite of all-cause death, non-fatal MI, and non-fatal stroke) at long-term follow-up; Aim 2) to evaluate the impact of CYP2C19 gene polymorphisms (loss of function alleles vs. non-loss of function alleles) on the risk of MALE (a composite of limb amputations, chronic threatening limb ischemia, acute limb ischemia, and limb revascularization) at long-term follow-up; and Aim 3) to evaluate the impact of CYP2C19 gene polymorphisms (loss of function alleles vs. non-loss of function alleles) on the risk of cerebrovascular events (CVE, a composite of any stroke and transient ischemic attack) at long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years with available CYP2C19 genotyping results obtained within the predefined period.

Exclusion Criteria:

* Absence of CYP2C19 genotyping results obtained within the predefined period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic atherosclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 5 years
  Defined as the composite of all-cause death, non-fatal MI, ornon-fatal stroke

SECONDARY OUTCOMES:
Major adverse limb events | 5 years
  A composite of limb amputations, chronic threatening limb ischemia, acute limb ischemia, or limb revascularization.
Net adverse clinical events | 5 years
  a composite of all-cause death, myocardial infarction, stroke, and major bleeding.
Cerebrovascular event | 5 years
  A composite of any stroke or transient ischemic attack.
Major bleeding | 5 years
  Defined in accordance with the Bleeding Academic research consortium as BARC type 3 to 5 bleeding.
Minor bleeding | 5 years
  Defined in accordance with the Bleeding Academic research consortium as BARC type 1 to 2 bleeding.
Clinically relevant bleeding | 5 years
  Defined in accordance with the Bleeding Academic research consortium as BARC type 2 to 5 bleeding.
Venous thromboembolic disease | 5 years
  Defined as the composite of deep vein thrombosis or pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UF Health, Gainesville, Florida
  - UF Health, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Result] Lee CR, Luzum JA, Sangkuhl K, Gammal RS, Sabatine MS, Stein CM, Kisor DF, Limdi NA, Lee YM, Scott SA, Hulot JS, Roden DM, Gaedigk A, Caudle KE, Klein TE, Johnson JA, Shuldiner AR. Clinical Pharmacogenetics Implementation Consortium Guideline for CYP2C19 Genotype and Clopidogrel Therapy: 2022 Update. Clin Pharmacol Ther. 2022 Nov;112(5):959-967. doi: 10.1002/cpt.2526. Epub 2022 Feb 8. PMID 35034351
- [Result] Angiolillo DJ, Capodanno D, Danchin N, Simon T, Bergmeijer TO, Ten Berg JM, Sibbing D, Price MJ. Derivation, Validation, and Prognostic Utility of a Prediction Rule for Nonresponse to Clopidogrel: The ABCD-GENE Score. JACC Cardiovasc Interv. 2020 Mar 9;13(5):606-617. doi: 10.1016/j.jcin.2020.01.226. PMID 32139218
- [Result] Pereira NL, Cresci S, Angiolillo DJ, Batchelor W, Capers Q 4th, Cavallari LH, Leifer D, Luzum JA, Roden DM, Stellos K, Turrise SL, Tuteja S; American Heart Association Professional/Public Education and Publications Committee of the Council on Genomic and Precision Medicine; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Peripheral Vascular Disease; and Stroke Council. CYP2C19 Genetic Testing for Oral P2Y12 Inhibitor Therapy: A Scientific Statement From the American Heart Association. Circulation. 2024 Aug 6;150(6):e129-e150. doi: 10.1161/CIR.0000000000001257. Epub 2024 Jun 20. PMID 38899464